CLINICAL TRIAL: NCT04626323
Title: Open, Randomized, Unicenter Study Comparing Metabolic Surgery With Intensive Medical Therapy to Treat Diabetic Kidney Disease
Brief Title: Randomized Study Comparing Metabolic Surgery With Intensive Medical Therapy to Treat Diabetic Kidney Disease
Acronym: OBESE-DKD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Responsible Party: Principal Investigator, Ricardo Vitor Cohen, MD, Ricardo Vitor Cohen, MD, PhD, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBESE-DKD; CAAE - 37013420500000070 (Other: Institutional Review Board)
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 2; Kidney Disease, Chronic; Kidney Injury
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity; Metabolic surgery; Gastric bypass; Diabetic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Diabetes Mellitus; Obesity; Diabetic Nephropathies | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: This will be an open-label, randomized trial involving sixty (60) patients with DKD and obesity who will undergo RYGB (intervention arm) or receive BMT (control arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB (intervention arm) (Experimental): Thirty (30) obese patients with DKD will undergo gastric bypass. Patients will also receive standard of care medical therapy for DKD (ACEI or ARB + SGLT2i) and T2DM (metformin, glitazones, incretin therapy - DPP4 inhibitor and GLP-1 analogs - and insulin, if necessary). Other comorbidities, such as hypertension and dyslipidemia, will be treated according to the latest recommendations of the ADA. The surgical procedure will consist of a laparoscopic surgery performed by an experienced surgeon (approximately 6000 bariatric surgeries), who is accredited as surgeon of excellence by the Brazilian Society of Bariatric and Metabolic Surgery and Surgical Review and Surgical Review Corporation program since 2009.
  Interventions: Procedure: Roux-en-Y gastric bypass; Drug: Best medical treatment
- BMT (control arm). (Active Comparator): Thirty (30) obese patients with DKD will undergo best medical treatment for DKD (ACEI or ARB + SGLT2i) and T2DM (metformin, glitazones, incretin therapy - DPP4 inhibitor and GLP-1 analogs - and insulin, if necessary). Other comorbidities, such as hypertension and dyslipidemia, will be treated according to the latest recommendations of the ADA.
  Interventions: Drug: Best medical treatment

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — 1. Pneumoperitoneum closed with Veress needle
  2. Identification of Treitz angle
  3. Measurement of biliary loop (50 cm)
  4. Bowel transection with linear stapler (white load)
  5. Measurement of the alimentary limb (100 cm)
  6. Laterolateral Entero-anastomoses (white load)
  7. Construction of gastric pouch distant about 3 cm from the esophageal-gastric junction with stomach section in the small curvature.
  8. Linear cutting anastomosis (gastrojejunostomy) from about 1 to 1.2 cm
  9. Anastomosis integrity evaluation by methylene blue test and/or perioperative air.
  Expected surgical time: 60 minutes
  Other Names: RYGB
  Arms: RYGB (intervention arm)
Drug: Best medical treatment — Patients will also receive standard of care medical therapy for DKD (ACEI or ARB + SGLT2i) and T2DM (metformin, glitazones, incretin therapy - DPP4 inhibitor and GLP-1 analogs - and insulin, if necessary).
  Other Names: BMT

SUMMARY:
Proven therapy for DKD is primarily limited to RAAS blockers and SLGT2i. Weight reduction has the potential to become an additional and much needed treatment option. Of all the weight reduction strategies metabolic surgery is suited to be the most effective. Yet no study has of yet compared the effect of metabolic surgery against best medical treatment on the progression of DKD. This pilot trial is designed to be the first determine the efficacy of metabolic surgery in slowing progression of DKD as compared to best medical therapy. The study design will address all the major limitations previously documented, including the major dilemma of estimating versus measuring GFR. Of note, the study's design will allow its sample size to be adjusted upward using an adaptive design if necessary, to achieve statistical significance. It will also inform study design and sample size issues for all future studies in this field. The payoff of establishing metabolic surgery as a new and effective intervention to slow progression to ESRD would be great in terms of reducing patient suffering and societal costs.

This will be an open-label, randomized trial involving sixty (60) patients with diabetic kidney disease (DKD) and obesity who will undergo Roux-en-Y gastric bypass (RYGB) in the intervention arm or receive best medical treatment (BMT) in the control arm.

The aim of this prospective, open, randomized study is to evaluate the efficacy and safety of RYGB surgery versus best medical treatment on the progression of DKD in patients with type 2 diabetes and obesity.

DETAILED DESCRIPTION:
This will be an open-label, randomized trial involving sixty (60) patients with DKD and obesity who will undergo RYGB (intervention arm) or receive BMT (control arm).

Thirty (30) obese patients with DKD will undergo gastric bypass. Patients will also receive standard of care medical therapy for DKD (ACEI or ARB + SGLT2i) and T2DM (metformin, glitazones, incretin therapy - DPP4 inhibitor and GLP-1 analogs - and insulin, if necessary). Other comorbidities, such as hypertension and dyslipidemia, will be treated according to the latest recommendations of the ADA. The surgical procedure will consist of a laparoscopic surgery performed by an experienced surgeon (approximately 6000 bariatric surgeries), who is accredited as surgeon of excellence by the Brazilian Society of Bariatric and Metabolic Surgery and Surgical Review and Surgical Review Corporation program since 2009.

Thirty (30) obese patients with DKD will undergo best medical treatment for DKD (ACEI or ARB + SGLT2i) and T2DM (metformin, glitazones, incretin therapy - DPP4 inhibitor and GLP-1 analogs - and insulin, if necessary). Other comorbidities, such as hypertension and dyslipidemia, will be treated according to the latest recommendations of the ADA.

Regarding medication therapy: Metformin will be maintained in the postoperative period while fasting glycemia is above 100 mg/dL unless contraindicated. Anti-antihypertensive drugs and medications for dyslipidemia will be maintained in the postoperative period, unless contraindicated. Micronutrient supplementation (vitamins and mineral salts) will be prescribed to all patients undergoing metabolic surgery. Patients allocated to the control group will receive the same supplementation if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥30 and ≤70 years
* Diabetic kidney disease as defined by an estimated glomerular filtration rate (eGFR) (as estimated by CKD-EPI creatinine + cystatin C equation)72 between 45-59l/min/1.73m2 and macroalbuminuria (≥ 300 mg/g) in a 24 hr urine sample
* BMI ≥30-40 kg/m2
* Fasting C-peptide over 1 ng/ml
* Negative glutamic acid decarboxylase autoantibodies test
* Patients having received accurate information about the surgery and requesting the procedure
* Patients having understood and accepted the need for long-term medical and surgical follow-up
* Effective method of contraception in women of child-bearing age
* Signed informed consent document

Exclusion Criteria:

* Refusal to participate
* Autoimmune diabetes/type 1 diabetes
* Previous abdominal operations that would complicate a metabolic surgery or increase surgical risk
* Previous malabsorptive and restrictive surgeries
* Malabsorptive syndromes and inflammatory bowel disease
* Significant and/or severe hepatic disease that may complicate metabolic surgery
* Pregnancy or women of childbearing age without effective contraceptive
* Recent history of neoplasia (< 5 years), except for non-melanoma skin neoplasms
* History of liver cirrhosis, active chronic hepatitis, active hepatitis B or hepatitis C
* Major cardiovascular event in the last 6 months
* Current angina
* Pulmonary embolism or severe thrombophlebitis in the last 2 years
* Positive HIV serum testing
* Mental incapacity or severe mental illness
* Severe psychiatric disorders that would complicate follow-up after randomization
* Alcoholism or illicit drug use
* Uncontrolled coagulopathy
* Participation in other clinical trials in the past 30 days
* Inability to tolerate RAAS blockers and/or SGLT2i
* Iodine allergy
* History of acute kidney injury requiring renal replacement therapy
* Dialysis dependency
* Kidney transplantation
* Use of immunosuppressive drugs, chemotherapy and/or radiotherapy
* Any disorder which, in the opinion of the investigator, might jeopardize subject's safety or compliance with the protocol

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean differenceGlomerular filtration rate (GFR) | At 12 and 36 months after randomization
  Mean difference in GFR between BMT and RYGB at the pre-specified time points of 12 and 36 months after randomization

SECONDARY OUTCOMES:
Change in twenty-four hour urinary albumin/protein excretion | From baseline to 12 and 36 months
  Change in 24h urinary albumin/protein excretion
Improvements in micro- or macroalbuminuria | From baseline to 12 and 36 months
  Proportion of patients who achieve improvements in micro- or macroalbuminuria from baseline to 12 and 36 months
Change in CKD stage and CKD prognostic risk | From baseline to 12 and 36 months
  Change in CKD stage and CKD prognostic risk from baseline to month 12 and 36
Change in GFR, eGFR and 24 hr creatinine clearance | From baseline to 12 and 36 months
  Change in GFR, eGFR and 24 hr creatinine clearance from baseline to months 12 and 36
Proportion of participants with ≥30%, ≥40%, and ≥50% reduction in GFR measurements | From baseline to 12 and 36 months
  Proportion of participants with ≥30%, ≥40%, and ≥50% reduction in GFR measurements (GFR, eGFR and 24 hr creatinine clearance) from baseline to months 12 and 36
Decline in eGFR, sustained low eGFR, kidney transplantation, maintenance dialysis, and kidney death | Time to occurrence (from baseline)
  Time to occurrence of sustained % decline in eGFR, sustained low eGFR, kidney transplantation, maintenance dialysis, and kidney death
Maintenance dialysis, kidney transplantation, kidney death, and GFR < 15 ml/min | At 12 and 36 months after randomization
  Individual and composite endpoints of maintenance dialysis, kidney transplantation, kidney death, and GFR < 15 ml/min at 12 and 36 months
Change in body weight | From baseline to 12 and 36 months
  Change in body weight from baseline to months 12 and 36
Change in body mass index | From baseline to 12 and 36 months
  Change in body mass index from baseline to months 12 and 36
Change in waist circumference | From baseline to 12 and 36 months
  Change in waist circumference from baseline to months 12 and 36
Medications to maintain optimal diabetes and blood pressure control | From baseline to 12 and 36 months
  Number and dose of medications to maintain optimal diabetes and blood pressure control from baseline to months 12 and 36
Change in fasting glucose | From baseline to 12 and 36 months
  Change in fasting glucose from baseline to months 12 and 36
Change in HbA1c | From baseline to 12 and 36 months
  Change in HbA1c from baseline to months 12 and 36
Change in basal insulin | From baseline to 12 and 36 months
  Change in basal insulin from baseline to months 12 and 36
Change in homeostasis model assessment (HOMA) scores | From baseline to 12 and 36 months
  Change in homeostasis model assessment (HOMA) scores from baseline to months 12 and 36
Remission in type 2 diabetes | At 12 and 36 months after randomization
  Achievement of partial or complete remission in type 2 diabetes by months 12 and 36
Change in blood pressure | From baseline to 12 and 36 months
  Change in blood pressure from baseline to months 12 and 36
Hypoglycemic adverse events | From baseline to 12 and 36 months
  Number of patients with confirmed or symptomatic hypoglycemic adverse events from baseline to months 12 and 36
Changes in total cholesterol, triglycerides, LDL and HDL levels | From baseline to 12 and 36 months
  Changes in total cholesterol, triglycerides, LDL and HDL levels from baseline to months 12 and 36
Number of participants achieving LDL < 100 mg/dL and HDL > 40mg/dL | From baseline to 12 and 36 months
  Number of participants achieving LDL < 100 mg/dL and HDL > 40mg/dL from baseline to months 12 and 36
Changes in serum calcium and phosphorus, | From baseline to 12 and 36 months
  Changes in serum calcium and phosphorus from baseline to months 12 and 36
Change in parathyroid hormone (PTH) | From baseline to 12 and 36 months
  Change in parathyroid hormone (PTH) from baseline to months 12 and 36
Change in mineral bone density | From baseline to 12 and 36 months
  Change in mineral bone density from baseline to months 12 and 36
Change in quality of life | From baseline to 12 and 36 months
  Change in quality of life measured by SF-36 questionnaire from baseline to months 12 and 36
Adverse events | From baseline to 12 and 36 months
  Number of patients with adverse events from baseline to months 12 and 36
Acute kidney injury | From baseline to 12 and 36 months
  Number of episodes of acute kidney injury from baseline to months 12 and 36
Adverse cardiovascular events (nonfatal stroke, nonfatal MI, cardiovascular death) | From baseline to 12 and 36 months
  Composite of major adverse cardiovascular events (nonfatal stroke, nonfatal MI, cardiovascular death) from baseline to months 12 and 36
Mortality | From baseline to 12 and 36 months
  Total mortality from baseline to months 12 and 36
Days hospitalized | From baseline to 12 and 36 months
  Number of days hospitalized from baseline to months 12 and 36
Change in urinary volume | From baseline to 12 and 36 months
  Change in urinary volume from baseline to months 12 and 36
Change in calcium and oxalate excretion | From baseline to 12 and 36 months
  Change in calcium and oxalate excretion from baseline to months 12 and 36
High sensitivity c-reactive protein | From baseline to 12 and 36 months
  Change in high sensitivity c-reactive protein from baseline to months 12 and 36
Change in muscle strength | From baseline to 12 and 36 months
  Change in muscle strength using one repetition maximum (1-RM) from baseline to months12 and 36
Kidney volumes | From baseline to 12 and 36 months
  Change in kidney volumes from baseline to months 12 and 36
Change in ventricular mass | From baseline to 12 and 36 months
  Change in left and right ventricular mass from baseline to months 12 and 36
Change in ejection fraction | From baseline to 12 and 36 months
  Change in left ventricular ejection fraction from baseline to months 12 and 36
Costs of care and health care utilization | From baseline to 12 and 36 months
  Costs of care and health care utilization from baseline to months 12 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo V Cohen, MD, PhD, Principal Investigator — Oswaldo Cruz German Hospital
Locations (1):
- Centro especializado em Obesidade e Diabetes do Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atkins RC, Zimmet P. Diabetic kidney disease: act now or pay later. Kidney Int. 2010 Mar;77(5):375-7. doi: 10.1038/ki.2009.509. No abstract available. PMID 20150934
- [Result] Mann JF, Gerstein HC, Pogue J, Bosch J, Yusuf S. Renal insufficiency as a predictor of cardiovascular outcomes and the impact of ramipril: the HOPE randomized trial. Ann Intern Med. 2001 Apr 17;134(8):629-36. doi: 10.7326/0003-4819-134-8-200104170-00007. PMID 11304102
- [Result] Afkarian M, Sachs MC, Kestenbaum B, Hirsch IB, Tuttle KR, Himmelfarb J, de Boer IH. Kidney disease and increased mortality risk in type 2 diabetes. J Am Soc Nephrol. 2013 Feb;24(2):302-8. doi: 10.1681/ASN.2012070718. Epub 2013 Jan 29. PMID 23362314
- [Result] Foley RN, Collins AJ. The growing economic burden of diabetic kidney disease. Curr Diab Rep. 2009 Dec;9(6):460-5. doi: 10.1007/s11892-009-0075-9. PMID 19954692
- [Result] (IHME) IfHMaE. Findings from the Global Burden of Disease Study 2017. Seattle, WA2018.
- [Result] World Health Organization Diabetes. 2018; https://www.who.int/news-room/fact-sheets/detail/diabetes.
- [Result] Alicic RZ, Rooney MT, Tuttle KR. Diabetic Kidney Disease: Challenges, Progress, and Possibilities. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2032-2045. doi: 10.2215/CJN.11491116. Epub 2017 May 18. PMID 28522654
- [Result] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S64-71. doi: 10.2337/dc12-s064. No abstract available. PMID 22187472
- [Result] Eckel RH, Kahn SE, Ferrannini E, Goldfine AB, Nathan DM, Schwartz MW, Smith RJ, Smith SR. Obesity and type 2 diabetes: what can be unified and what needs to be individualized? J Clin Endocrinol Metab. 2011 Jun;96(6):1654-63. doi: 10.1210/jc.2011-0585. PMID 21602457
- [Result] Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S; RENAAL Study Investigators. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med. 2001 Sep 20;345(12):861-9. doi: 10.1056/NEJMoa011161. PMID 11565518
- [Result] Lewis EJ, Hunsicker LG, Clarke WR, Berl T, Pohl MA, Lewis JB, Ritz E, Atkins RC, Rohde R, Raz I; Collaborative Study Group. Renoprotective effect of the angiotensin-receptor antagonist irbesartan in patients with nephropathy due to type 2 diabetes. N Engl J Med. 2001 Sep 20;345(12):851-60. doi: 10.1056/NEJMoa011303. PMID 11565517
- [Result] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Result] de Boer IH, Rue TC, Hall YN, Heagerty PJ, Weiss NS, Himmelfarb J. Temporal trends in the prevalence of diabetic kidney disease in the United States. JAMA. 2011 Jun 22;305(24):2532-9. doi: 10.1001/jama.2011.861. PMID 21693741
- [Result] Friedman AN, Wolfe B. Is Bariatric Surgery an Effective Treatment for Type II Diabetic Kidney Disease? Clin J Am Soc Nephrol. 2016 Mar 7;11(3):528-35. doi: 10.2215/CJN.07670715. Epub 2015 Oct 8. PMID 26450931
- [Result] Friedman AN, Moe S, Fadel WF, Inman M, Mattar SG, Shihabi Z, Quinney SK. Predicting the glomerular filtration rate in bariatric surgery patients. Am J Nephrol. 2014;39(1):8-15. doi: 10.1159/000357231. Epub 2013 Dec 19. PMID 24356416
- [Result] Foster MC, Hwang SJ, Porter SA, Massaro JM, Hoffmann U, Fox CS. Fatty kidney, hypertension, and chronic kidney disease: the Framingham Heart Study. Hypertension. 2011 Nov;58(5):784-90. doi: 10.1161/HYPERTENSIONAHA.111.175315. Epub 2011 Sep 19. PMID 21931075
- [Result] Wiggins JE, Goyal M, Sanden SK, Wharram BL, Shedden KA, Misek DE, Kuick RD, Wiggins RC. Podocyte hypertrophy, "adaptation," and "decompensation" associated with glomerular enlargement and glomerulosclerosis in the aging rat: prevention by calorie restriction. J Am Soc Nephrol. 2005 Oct;16(10):2953-66. doi: 10.1681/ASN.2005050488. Epub 2005 Aug 24. PMID 16120818
- [Result] D'Agati VD, Chagnac A, de Vries AP, Levi M, Porrini E, Herman-Edelstein M, Praga M. Obesity-related glomerulopathy: clinical and pathologic characteristics and pathogenesis. Nat Rev Nephrol. 2016 Aug;12(8):453-71. doi: 10.1038/nrneph.2016.75. Epub 2016 Jun 6. PMID 27263398
- [Result] Stern JS, Gades MD, Wheeldon CM, Borchers AT. Calorie restriction in obesity: prevention of kidney disease in rodents. J Nutr. 2001 Mar;131(3):913S-917S. doi: 10.1093/jn/131.3.913S. PMID 11238785
- [Result] Nangaku M, Izuhara Y, Usuda N, Inagi R, Shibata T, Sugiyama S, Kurokawa K, van Ypersele de Strihou C, Miyata T. In a type 2 diabetic nephropathy rat model, the improvement of obesity by a low calorie diet reduces oxidative/carbonyl stress and prevents diabetic nephropathy. Nephrol Dial Transplant. 2005 Dec;20(12):2661-9. doi: 10.1093/ndt/gfi096. Epub 2005 Sep 27. PMID 16188903
- [Result] Ohtomo S, Izuhara Y, Nangaku M, Dan T, Ito S, van Ypersele de Strihou C, Miyata T. Body weight control by a high-carbohydrate/low-fat diet slows the progression of diabetic kidney damage in an obese, hypertensive, type 2 diabetic rat model. J Obes. 2010;2010:136502. doi: 10.1155/2010/136502. Epub 2010 Feb 17. PMID 20700413
- [Result] Gugliucci A, Kotani K, Taing J, Matsuoka Y, Sano Y, Yoshimura M, Egawa K, Horikawa C, Kitagawa Y, Kiso Y, Kimura S, Sakane N. Short-term low calorie diet intervention reduces serum advanced glycation end products in healthy overweight or obese adults. Ann Nutr Metab. 2009;54(3):197-201. doi: 10.1159/000217817. Epub 2009 May 6. PMID 19420913
- [Result] Wycherley TP, Brinkworth GD, Noakes M, Buckley JD, Clifton PM. Effect of caloric restriction with and without exercise training on oxidative stress and endothelial function in obese subjects with type 2 diabetes. Diabetes Obes Metab. 2008 Nov;10(11):1062-73. doi: 10.1111/j.1463-1326.2008.00863.x. Epub 2008 Apr 22. PMID 18435772
- [Result] Seshadri P, Iqbal N, Stern L, Williams M, Chicano KL, Daily DA, McGrory J, Gracely EJ, Rader DJ, Samaha FF. A randomized study comparing the effects of a low-carbohydrate diet and a conventional diet on lipoprotein subfractions and C-reactive protein levels in patients with severe obesity. Am J Med. 2004 Sep 15;117(6):398-405. doi: 10.1016/j.amjmed.2004.04.009. PMID 15380496
- [Result] Tuck ML, Sowers J, Dornfeld L, Kledzik G, Maxwell M. The effect of weight reduction on blood pressure, plasma renin activity, and plasma aldosterone levels in obese patients. N Engl J Med. 1981 Apr 16;304(16):930-3. doi: 10.1056/NEJM198104163041602. PMID 7010165
- [Result] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Result] Laferrere B, Teixeira J, McGinty J, Tran H, Egger JR, Colarusso A, Kovack B, Bawa B, Koshy N, Lee H, Yapp K, Olivan B. Effect of weight loss by gastric bypass surgery versus hypocaloric diet on glucose and incretin levels in patients with type 2 diabetes. J Clin Endocrinol Metab. 2008 Jul;93(7):2479-85. doi: 10.1210/jc.2007-2851. Epub 2008 Apr 22. PMID 18430778
- [Result] Gregg EW, Chen H, Wagenknecht LE, Clark JM, Delahanty LM, Bantle J, Pownall HJ, Johnson KC, Safford MM, Kitabchi AE, Pi-Sunyer FX, Wing RR, Bertoni AG; Look AHEAD Research Group. Association of an intensive lifestyle intervention with remission of type 2 diabetes. JAMA. 2012 Dec 19;308(23):2489-96. doi: 10.1001/jama.2012.67929. PMID 23288372
- [Result] UK Prospective Diabetes Study (UKPDS). X. Urinary albumin excretion over 3 years in diet-treated type 2, (non-insulin-dependent) diabetic patients, and association with hypertension, hyperglycaemia and hypertriglyceridaemia. Diabetologia. 1993 Oct;36(10):1021-9. PMID 8243850
- [Result] Heshka S, Anderson JW, Atkinson RL, Greenway FL, Hill JO, Phinney SD, Kolotkin RL, Miller-Kovach K, Pi-Sunyer FX. Weight loss with self-help compared with a structured commercial program: a randomized trial. JAMA. 2003 Apr 9;289(14):1792-8. doi: 10.1001/jama.289.14.1792. PMID 12684357
- [Result] Dansinger ML, Gleason JA, Griffith JL, Selker HP, Schaefer EJ. Comparison of the Atkins, Ornish, Weight Watchers, and Zone diets for weight loss and heart disease risk reduction: a randomized trial. JAMA. 2005 Jan 5;293(1):43-53. doi: 10.1001/jama.293.1.43. PMID 15632335
- [Result] Schiavon CA, Bersch-Ferreira AC, Santucci EV, Oliveira JD, Torreglosa CR, Bueno PT, Frayha JC, Santos RN, Damiani LP, Noujaim PM, Halpern H, Monteiro FLJ, Cohen RV, Uchoa CH, de Souza MG, Amodeo C, Bortolotto L, Ikeoka D, Drager LF, Cavalcanti AB, Berwanger O. Effects of Bariatric Surgery in Obese Patients With Hypertension: The GATEWAY Randomized Trial (Gastric Bypass to Treat Obese Patients With Steady Hypertension). Circulation. 2018 Mar 13;137(11):1132-1142. doi: 10.1161/CIRCULATIONAHA.117.032130. Epub 2017 Nov 13. PMID 29133606
- [Result] Scheurlen KM, Probst P, Kopf S, Nawroth PP, Billeter AT, Muller-Stich BP. Metabolic surgery improves renal injury independent of weight loss: a meta-analysis. Surg Obes Relat Dis. 2019 Jun;15(6):1006-1020. doi: 10.1016/j.soard.2019.03.013. Epub 2019 Mar 20. PMID 31104957
- [Result] Peromaa-Haavisto P, Tuomilehto H, Kossi J, Virtanen J, Luostarinen M, Pihlajamaki J, Kakela P, Victorzon M. Obstructive sleep apnea: the effect of bariatric surgery after 12 months. A prospective multicenter trial. Sleep Med. 2017 Jul;35:85-90. doi: 10.1016/j.sleep.2016.12.017. Epub 2017 Jan 12. PMID 28549834
- [Result] Le Jemtel TH, Samson R, Jaiswal A, Lewine EB, Oparil S. Regression of Left Ventricular Mass After Bariatric Surgery. Curr Hypertens Rep. 2017 Sep;19(9):68. doi: 10.1007/s11906-017-0767-5. PMID 28755274
- [Result] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Result] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Aminian A, Brethauer SA, Navaneethan SD, Singh RP, Pothier CE, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric Surgery versus Intensive Medical Therapy for Diabetes - 5-Year Outcomes. N Engl J Med. 2017 Feb 16;376(7):641-651. doi: 10.1056/NEJMoa1600869. PMID 28199805
- [Result] Muller-Stich BP, Senft JD, Warschkow R, Kenngott HG, Billeter AT, Vit G, Helfert S, Diener MK, Fischer L, Buchler MW, Nawroth PP. Surgical versus medical treatment of type 2 diabetes mellitus in nonseverely obese patients: a systematic review and meta-analysis. Ann Surg. 2015 Mar;261(3):421-9. doi: 10.1097/SLA.0000000000001014. PMID 25405560
- [Result] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Result] Neff KJ, Elliott JA, Corteville C, Abegg K, Boza C, Lutz TA, Docherty NG, le Roux CW. Effect of Roux-en-Y gastric bypass and diet-induced weight loss on diabetic kidney disease in the Zucker diabetic fatty rat. Surg Obes Relat Dis. 2017 Jan;13(1):21-27. doi: 10.1016/j.soard.2016.08.026. Epub 2016 Aug 18. PMID 27665150
- [Result] Canney AL, Cohen RV, Elliott JA, M Aboud C, Martin WP, Docherty NG, le Roux CW. Improvements in diabetic albuminuria and podocyte differentiation following Roux-en-Y gastric bypass surgery. Diab Vasc Dis Res. 2020 Jan-Feb;17(1):1479164119879039. doi: 10.1177/1479164119879039. Epub 2019 Nov 14. PMID 31726864
- [Result] O'Brien R, Johnson E, Haneuse S, Coleman KJ, O'Connor PJ, Fisher DP, Sidney S, Bogart A, Theis MK, Anau J, Schroeder EB, Arterburn D. Microvascular Outcomes in Patients With Diabetes After Bariatric Surgery Versus Usual Care: A Matched Cohort Study. Ann Intern Med. 2018 Sep 4;169(5):300-310. doi: 10.7326/M17-2383. Epub 2018 Aug 7. PMID 30083761
- [Result] Young L, Nor Hanipah Z, Brethauer SA, Schauer PR, Aminian A. Long-term impact of bariatric surgery in diabetic nephropathy. Surg Endosc. 2019 May;33(5):1654-1660. doi: 10.1007/s00464-018-6458-8. Epub 2018 Sep 24. PMID 30251143
- [Result] Shulman A, Peltonen M, Sjostrom CD, Andersson-Assarsson JC, Taube M, Sjoholm K, le Roux CW, Carlsson LMS, Svensson PA. Incidence of end-stage renal disease following bariatric surgery in the Swedish Obese Subjects Study. Int J Obes (Lond). 2018 Jun;42(5):964-973. doi: 10.1038/s41366-018-0045-x. Epub 2018 Feb 26. PMID 29568103
- [Result] Friedman AN, Wang J, Wahed AS, Docherty NG, Fennern E, Pomp A, Purnell JQ, le Roux CW, Wolfe B. The Association Between Kidney Disease and Diabetes Remission in Bariatric Surgery Patients With Type 2 Diabetes. Am J Kidney Dis. 2019 Dec;74(6):761-770. doi: 10.1053/j.ajkd.2019.05.013. Epub 2019 Jul 19. PMID 31331758
- [Result] Inge TH, Laffel LM, Jenkins TM, Marcus MD, Leibel NI, Brandt ML, Haymond M, Urbina EM, Dolan LM, Zeitler PS; Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) and Treatment Options of Type 2 Diabetes in Adolescents and Youth (TODAY) Consortia. Comparison of Surgical and Medical Therapy for Type 2 Diabetes in Severely Obese Adolescents. JAMA Pediatr. 2018 May 1;172(5):452-460. doi: 10.1001/jamapediatrics.2017.5763. PMID 29532078
- [Result] Imam TH, Fischer H, Jing B, Burchette R, Henry S, DeRose SF, Coleman KJ. Estimated GFR Before and After Bariatric Surgery in CKD. Am J Kidney Dis. 2017 Mar;69(3):380-388. doi: 10.1053/j.ajkd.2016.09.020. Epub 2016 Dec 4. PMID 27927587
- [Result] Friedman AN, Wahed AS, Wang J, Courcoulas AP, Dakin G, Hinojosa MW, Kimmel PL, Mitchell JE, Pomp A, Pories WJ, Purnell JQ, le Roux C, Spaniolas K, Steffen KJ, Thirlby R, Wolfe B. Effect of Bariatric Surgery on CKD Risk. J Am Soc Nephrol. 2018 Apr;29(4):1289-1300. doi: 10.1681/ASN.2017060707. Epub 2018 Jan 15. PMID 29335242
- [Result] Aminian A, Brethauer SA, Kirwan JP, Kashyap SR, Burguera B, Schauer PR. How safe is metabolic/diabetes surgery? Diabetes Obes Metab. 2015 Feb;17(2):198-201. doi: 10.1111/dom.12405. Epub 2014 Nov 19. PMID 25352176
- [Result] Cohen JB, Tewksbury CM, Torres Landa S, Williams NN, Dumon KR. National Postoperative Bariatric Surgery Outcomes in Patients with Chronic Kidney Disease and End-Stage Kidney Disease. Obes Surg. 2019 Mar;29(3):975-982. doi: 10.1007/s11695-018-3604-2. PMID 30443719
- [Result] Nasr SH, D'Agati VD, Said SM, Stokes MB, Largoza MV, Radhakrishnan J, Markowitz GS. Oxalate nephropathy complicating Roux-en-Y Gastric Bypass: an underrecognized cause of irreversible renal failure. Clin J Am Soc Nephrol. 2008 Nov;3(6):1676-83. doi: 10.2215/CJN.02940608. Epub 2008 Aug 13. PMID 18701613
- [Result] Sundbom M, Naslund E, Vidarsson B, Thorell A, Ottoson J. Low overall mortality during 10 years of bariatric surgery: nationwide study on 63,469 procedures from the Scandinavian Obesity Registry. Surg Obes Relat Dis. 2020 Jan;16(1):65-70. doi: 10.1016/j.soard.2019.10.012. Epub 2019 Oct 21. PMID 31753796
- [Result] Cummings DE, Cohen RV. Bariatric/Metabolic Surgery to Treat Type 2 Diabetes in Patients With a BMI <35 kg/m2. Diabetes Care. 2016 Jun;39(6):924-33. doi: 10.2337/dc16-0350. PMID 27222550
- [Result] Batterham RL, Cummings DE. Mechanisms of Diabetes Improvement Following Bariatric/Metabolic Surgery. Diabetes Care. 2016 Jun;39(6):893-901. doi: 10.2337/dc16-0145. PMID 27222547
- [Result] Cohen RV, Shikora S, Petry T, Caravatto PP, Le Roux CW. The Diabetes Surgery Summit II Guidelines: a Disease-Based Clinical Recommendation. Obes Surg. 2016 Aug;26(8):1989-91. doi: 10.1007/s11695-016-2237-6. PMID 27189354
- [Result] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Nanni G, Castagneto M, Bornstein S, Rubino F. Bariatric-metabolic surgery versus conventional medical treatment in obese patients with type 2 diabetes: 5 year follow-up of an open-label, single-centre, randomised controlled trial. Lancet. 2015 Sep 5;386(9997):964-73. doi: 10.1016/S0140-6736(15)00075-6. PMID 26369473
- [Result] Cohen RV, Pinheiro JC, Schiavon CA, Salles JE, Wajchenberg BL, Cummings DE. Effects of gastric bypass surgery in patients with type 2 diabetes and only mild obesity. Diabetes Care. 2012 Jul;35(7):1420-8. doi: 10.2337/dc11-2289. PMID 22723580
- [Result] Navaneethan SD, Yehnert H, Moustarah F, Schreiber MJ, Schauer PR, Beddhu S. Weight loss interventions in chronic kidney disease: a systematic review and meta-analysis. Clin J Am Soc Nephrol. 2009 Oct;4(10):1565-74. doi: 10.2215/CJN.02250409. Epub 2009 Sep 17. PMID 19808241
- [Result] Cohen RV, Pereira TV, Aboud CM, Caravatto PP, Petry TB, Correa JL, Schiavon CA, Correa M, Pompilio CE, Pechy FN, le Roux CW; MOMS Study Investigators. Microvascular Outcomes after Metabolic Surgery (MOMS) in patients with type 2 diabetes mellitus and class I obesity: rationale and design for a randomised controlled trial. BMJ Open. 2017 Jan 11;7(1):e013574. doi: 10.1136/bmjopen-2016-013574. PMID 28077412
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Friedman AN, Chang AR, Chuah LL, Favre GA, Grangeon-Chapon C, Lane KA, Li Y, le Roux CW, Lieske JC, Morales E, Porrini E, Chagnac A. Measurement, Estimation, and Correlates of the GFR before and after Bariatric Surgery. J Am Soc Nephrol. 2026 Jan 1;37(1):110-119. doi: 10.1681/ASN.0000000797. Epub 2025 Jul 15. PMID 40663401
- See also: Obesity and Diabetes Center — https://centrodeobesidadeediabetes.org.br/
- See also: Oswaldo Cruz German Hospital — https://www.hospitaloswaldocruz.org.br/